CLINICAL TRIAL: NCT04773626
Title: Evaluation of the Role of Tumor Deposits on the Prognosis of Colorectal Carcinoma
Brief Title: Tumor Deposits in Cancer Colon
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Fathi Mosa, Resident doctor, Assiut University
Other Study IDs: Not yet
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Cancer of Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assessment of correlation between tumor deposits and clinicopathological characteristics of colorectal cancer.
2. Detection of association between tumor deposits and stage of colorectal cancer.
3. Evaluate the relationship between tumor deposits and prognosis of colorectal cancer patient.

DETAILED DESCRIPTION:
Colorectal cancer remains the third most common cancer and the third leading cause of cancer-related deaths. For colon cancer alone, 101,220 new cases were projected to occur in 2019, causing51,020 deaths.

A number of risk factors have been identified that influence susceptibility to colorectal cancer, including a family history, the presence of adenomatous polyps, inflammatory bowel disease (ulcerative colitis or Crohn's disease), and number of environmental factors of which diet is the most significant.

CRC differs from many other cancers in that diagnosis of the disease can be made earlier by screening techniques including colonoscopy. The progression of CRC is well established and begins with hyperproliferation of the colonic mucosa and adenoma formation and then adenocarcinomas that vary in metastatic potential.

The progression from normal intestinal epithelium to an invasive carcinoma is estimated to take 7-12 years. With the advent of early screening measures developed over the last few decades, CRC has become a preventable disease by treating patients with adenomatous polyps. Nearly 50% of patients diagnosed with CRC develop metastasis within five years. Most commonly these tumors metastasize to the liver and lungs but may be discovered in many other sites.

Despite significant improvements in both prevention and screening over the last twenty years, about 36,500 (36%) of such cases are still being diagnosed in stage III, with regional lymph node involvement (LN+, N1a-b, N2a-b) or tumor deposits (TD+, N1c).

Tumor deposits (TDs) or mesenteric tumor satellites were firs described in rectal carcinoma by Gabriel et al at St. Mark's Hospital in 1935. Subsequently, TDs have been detected in various malignancies other than colorectal carcinoma, including gastric, pancreatic, gallbladder, and bile duct carcinomas . Over the years, there is much debate about the genesis, histopathologic characteristics, and prognostic value of TDs.

TDs are associated with advanced colorectal carcinoma stage and poor prognosis, with variable outcome due to different definitions of TDs.

Before the 5th edition, published in 1997, TNM classification did not consider microscopic TDs to be lymph node metastases (LNMs), and they classified them as discontinuous extension in the T category .

In the 5th TNM edition the 3-mm rule was introduced, which stated that TDs >3mm in diameter were LNMs .

In the 6th edition published in 2002, TDs were classified based on the contour of the deposit. A TD with a smooth contour was considered as LMN, whereas a TD with an irregular contour was considered as venous invasion (V1/2) or lymphatic invasion (L1).

The 8th TNM Edition clarified that the presence of TDs does not change the primary tumor T category, but changes the node status (N) to pN1c if all regional lymph nodes are negative on pathological examination.

In studies of rectal cancer patients, it should be taken into account that TDs may indicate microscopic residuals of the main tumor after neoadjuvant chemo radiation and not discontinuous foci of tumor as indicated in the classic definition of TDs.

The presence of TDs was an independent adverse prognostic factor that was significantly associated with shorter disease-free survival independent of lymph node status in stage IV colorectal cancer patients who underwent simultaneous resection for synchronous colorectal liver metastases.

After chemo-radiotherapy, rectal cancer is usually associated with small clusters of tumor cells or isolated tumor cells, scattered within or outside the rectal wall which are often associated to fibrosis and chronic inflammation, as well as other radiation induced changes. The prognostic significance of TDs in rectal adenocarcinoma following neoadjuvant chemoradiation has not yet been determined, although this remains an important issue given that patients who receive neoadjuvant chemoradiation have more advanced tumors and the highest risk of distant and local recurrences.

TDs were associated with higher rates of lymph node involvement, distant metastases and reduced survival; more over TDs are associated with aggressive characteristics, including higher rates of positive circumferential resection margins.

ELIGIBILITY:
Inclusion Criteria:

- 1-This retrospective study includes primary invasive colorectal carcinoma samples from Egyptian patients.

2-Patients who underwent resection of colorectal cancer will be included in our study.

Exclusion Criteria:

* 1-All patients who underwent endoscopic biopsies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. This retrospective study includes primary invasive colorectal carcinoma samples from Egyptian patients that will be retrieved from the registry of Pathology department, South Egypt Cancer Institute and Assiut University Hospital.
  2. All patients who underwent resection of colorectal cancer will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the relationship between tumor deposits and prognosis of colorectal cancer patient. | 2 years
  1. Assessment of correlation between tumor deposits and clinicopathological characteristics of colorectal cancer.
  2. Detection of correlation between tumor deposits and stage of colorectal cancer.
  3. Correlation between tumor deposits and prognosis of colorectal cancer, clinicopathological characteristics of colorectal cancer, stage of colorectal cancer".

REFERENCES:
- [Background] Peparini N. Beyond T, N and M: The impact of tumor deposits on the staging and treatment of colorectal and gastric carcinoma. Surg Oncol. 2018 Jun;27(2):129-137. doi: 10.1016/j.suronc.2018.02.007. Epub 2018 Feb 21. PMID 29937162